CLINICAL TRIAL: NCT05656105
Title: PET Imaging of Neuroinflammation in Patients With Neurological Dysfunction After SARS-CoV-2 Infection
Brief Title: Positron Emission Tomography (PET) Imaging of Neuroinflammation in Patients With Neurological Dysfunction After Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV 2) Infection
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R22-209
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: SARS CoV-2 Post-Acute Sequelae

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healty Volunteers (Experimental)
  Interventions: Drug: DPA-714 PET/MRI
- PASC (Experimental): Patients meeting the case definition criteria for PASC
  Interventions: Drug: DPA-714 PET/MRI

INTERVENTIONS:
Drug: DPA-714 PET/MRI — DPA-714 PET/MRI

SUMMARY:
This clinical imaging study will use the small molecule translocator protein (TSPO) ligand, Fluorodeoxyglucose(18F)-labeled DPA-714, to visualize and quantify neuroinflammation in individuals with post-acute sequelae of SARS-CoV-2 (PASC) . The brain uptake of DPA-714 will be contrasted with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age
2. Healthy volunteer OR Clinical diagnosis of post-acute sequelae of SARS-CoV-2 (PASC)
3. High or mixed affinity binder for TSPO ligands based on genotyping for single nucleotide polymorphism (SNP) rs6971.
4. PASC participants must have been previously infected with SARS-CoV-2. Their neurological symptoms must have been present for at least four weeks prior to the enrollment.
5. Healthy control participants must have no neurological symptoms

Exclusion Criteria:

1. Contraindication to MRI
2. Pregnancy
3. Lactation
4. Individuals who are unable to participate in the imaging portion due to severity of their medical condition
5. Chronic infectious disease (e.g. HIV, HCV)
6. Viral or bacterial illness requiring medical attention and/or antibiotics within 1 month of study participation
7. Diagnosis of cancer, including leukemia
8. Blood or blood clotting disorder
9. Except for individuals with Multiple Sclerosis (MS), a diagnosis of autoimmune disease is exclusionary
10. Positive urine β-hCG test day of procedure or a serum human chorionic gonadotropin (hCG) test within 48 hours prior to the administration of [18F]DPA-714.11.

11Currently enrolled in a clinical trial utilizing experimental therapies. 12. Currently taking experimental therapies 13. Low affinity binder for TSPO ligands based on genotyping for SNP rs6971.

The following exclusionary criteria apply only to PASC patients and healthy controls:

14. Self-reported history of moderate or severe traumatic brain injury 15. Self-reported history of whiplash injury 16. Self-reported history of Inflammatory bowel disease (IBD). (Individuals with Irritable Bowel Syndrome (IBS) and no signs of inflammation will be allowed to participate.) 17. The following blood test results (at screening) will be exclusionary: 18. Rheumatoid Factor (RF) => 14 IntUnits/mL, 19. Anti-nuclear antibody (ANA) > 1:80, 20. Erythrocyte sedimentation rate (ESR) > 60mm/hour, 21.High sensitivity C-reactive protein (hsCRP) > 10mg/L, 22. Complete blood count (CBC) results indicating acute infection, anemia, or other condition, 23. T3, T4, or thyroid-stimulating hormone (TSH) levels out of normal range, 24. Fasting glucose > 100 mg/dL, 25. Blood chemistry results indicating organ damage or other serious medical condition 26. Use of illicit substances within the past 6 months 27. Self-reported diagnosis of Type I or Type II diabetes 28. Healthy controls must not regularly take over-the-counter anti-inflammatory medication, analgesics (except aspirin), or sleep medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of regional brain TSPO levels using PET in participants with neurological PASC and healthy volunteers | Injection/scan date to clinical follow-up. (Usually within 6 weeks)
  PET measures of TSPO binding in brain regions including cerebral cortex, thalami, and brainstem will be quantified in symptomatic study participants and healthy volunteers will be collected and compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No